CLINICAL TRIAL: NCT03859895
Title: Zoledronate In the Prevention of Paget's Disease: Long Term Extension
Acronym: ZiPP-LTE
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor
Other Study IDs: AC18051; 245197 (Other: IRAS (Integrated Research Application System)); 18/ES/0086 (Other: Research Ethics Committee (EoSRES))
Record Dates: First submitted 2019-01-31; First posted 2019-03-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Paget Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, saliva samples and stool samples will be collected from participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational (without bone scan): Former Observational Arm participants of the ZiPP trial.
- Observational (with bone scan): Former Interventional Arm participants of the ZiPP trial.

SUMMARY:
Paget's disease of the bone (PDB) is a metabolic bone disorder which in some individuals can cause pain, bone deformity, arthritis and deafness, although in many patients it does not cause symptoms. Paget's disease has a strong genetic component and SQSTM1 is the most important susceptibility gene. People who inherit mutations in SQSTM1 have a high risk of developing PDB later in life. This study is an extension of the ZiPP (Zoledronate in the Prevention of Paget's) study which was is randomised trial currently in progress to determine if the bisphosphonate zoledronic acid (ZA) can prevent or delay the development of PDB-like bone lesions compared with a dummy treatment (placebo) in people who inherit SQSMT1 gene mutations. Although the ZiPP study will provide information on whether early ZA treatment can favourably influence bone lesion development the significance of this to the patient in terms of symptoms is unclear as yet. The aim of the extension study is to keep these individuals under surveillance for any symptoms or signs of PDB over a further 5 year period and to evaluate if there has been any progression of PDB-like lesions by bone scan at the end of this period.

DETAILED DESCRIPTION:
It is at present unclear whether intervention with bisphosphonates is of clinical benefit in early PDB. Although the ZiPP study is expected to provide information on whether ZA can favourably influence the development of bone lesions characteristic of early PDB as determined by radionuclide bone scan imaging, longer term follow up is required to determine if this will translate into clinical benefit. The extension study described here will provide new information on the natural history of PDB by follow up of people that took part in the ZIPP trial. Although the ZIPP-LTE study is an observational study, treatment for PDB may be given to participants according to normal clinical practice if they develop signs or symptoms of PDB during the extension. Treatment will therefore be offered to all participants that develop symptoms of PDB during follow up. Additionally, subjects that were previously been exposed to ZA in the core study will also be offered further ZA or another bisphosphonate licensed for PDB if they develop evidence of increased metabolic activity thought to be due to PDB, even if asymptomatic. The reason for this is that adverse effects are rare in patients who have previously been treated with ZA but are common on first exposure to ZA. Both therapeutic approaches are commonly used in patients with early PDB with no evidence that one is superior to another. In addition to providing information on the natural history of PDB, part of the aim of the extension will be to evaluate the risks and benefits of these two approaches to standard care of in terms of new lesion development, pain, quality of life and adverse events in the context of people who inherit SQSTM1 mutations.

ELIGIBILITY:
Inclusion Criteria:

* Subject that participated in ZiPP
* Participant willing and able to consent and comply with the study protocol.

Exclusion Criteria:

* Unable or unwilling to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients recruited to the ZiPP Trial (2008-005667-34)
Sampling Method: Non-Probability Sample
Enrollment: 287 (Estimated)
Dates: Start 2019-04-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint (former ZiPP interventional arm): The proportion of patients that develop PDB-like bone lesions | 5 year time-point
  The proportion of patients in each of the randomisation groups that develop PDB-like bone lesions by the end of study assessed by radionuclide bone scan.
Primary Endpoint (former ZiPP observational arm): proportion of individuals that develop abnormalities suggestive of PDB | During follow-up period
  The primary endpoint will be to evaluate the proportion of individuals that develop biochemical or clinical abnormalities suggestive of PDB over a the 10-year duration of follow up.

SECONDARY OUTCOMES:
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to the number of new bone lesions assessed by radionuclide bone scan. | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Evaluate differences between ZiPP treatment and placebo groups for change in bone lesion activity by semi-quantitative analysis of radionuclide bone scans (method described by Patel et al (1995)). | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to SF36 (36-Item Short Form Survey) scores. | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to HAQ (Health Assessment Questionnaire) scores. | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to EQ5D (EuroQol five dimension scale) scores. | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to IPAQ (International Physical Activity Questionnaire) scores. | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to BPI (Brief Pain Inventory Scale) scores. | 5 year time-point
Secondary Endpoint (former ZiPP interventional arm): Differences between ZiPP trial treatment and placebo groups with regard to development of PDB-related skeletal events (PRSE). | 5 year time-point
  Defined as new bone lesions thought to be due to PDB on imaging OR complications of PDB such as pathological fractures, bone deformity, deafness, and joint replacement surgery OR administration of treatment for PDB because of pain localised to an affected site in a patient with metabolically active disease.
Secondary Endpoint (former ZiPP observational arm): Health-related quality of life in ZiPP trial observational arm participants assessed using EQ5D. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Health-related quality of life in ZiPP trial observational arm participants assessed using SF36. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Health-related quality of life in ZiPP trial observational arm participants assessed using BPI. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Health-related quality of life in ZiPP trial observational arm participants assessed using HAQ. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Health-related quality of life in ZiPP trial observational arm participants assessed using IPAQ. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Pain in ZiPP trial observational arm participants assessed using EQ5D. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Pain in ZiPP trial observational arm participants assessed using SF36. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Pain in ZiPP trial observational arm participants assessed using BPI. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Anxiety in ZiPP trial observational arm participants assessed using EQ5D. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Anxiety in ZiPP trial observational arm participants assessed using SF36. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Depression in ZiPP trial observational arm participants assessed using SF-36. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Depression in ZiPP trial observational arm participants assessed using BPI. | 5 year time-point
Secondary Endpoint (former ZiPP observational arm): Depression in ZiPP trial observational arm participants assessed using EQ5D. | 5 year time-point

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Ralston, Prof, Principal Investigator — Univeristy of Edinburgh
Locations (21):
- Australia (5):
  - University Hospital Geelong, Geelong
  - Sir Charles Gardner Hospital, Nedlands
  - Royal Newcastle Centre, Newcastle
  - University of Sydney, Sydney
  - University of Queensland, Toowoomba
- University Hospital Saint-Luc, Brussels, Belgium
- St. Vincent's University Hospital, Dublin, Ireland
- Italy (3):
  - University Hospital of Careggi, Florence
  - University of Siena, Siena
  - University of Turin, Turin
- New Zealand (2):
  - University of Auckland, Auckland
  - The Princess Margaret Hospital, Christchurch
- Spain (2):
  - Univeristy of Barcelona, Barcelona
  - University Hospital of Salamanca, Salamanca
- United Kingdom (7):
  - University of Bristol, Bristol, England
  - University of Liverpool, Liverpool, England
  - Guy's and St Thomas Hospital NHS Trust, London, England
  - King's College Hospital, London, England
  - Manchester Royal Infirmary, Manchester, England
  - NHS Lothian, Edinburgh, Scotland
  - Wrexham Maelor Hospital, Wrexham, Wales

IPD SHARING:
Plan to Share IPD: Undecided